

## Consent form

Title of Project: Continuous Glucose Monitoring: An evaluation of impact on improving the efficiency of diagnostic processes and enhancing patient safety in the management of reactive and spontaneous hypoglycaemia.

**IRAS ID 265405** 

REC ref 19/LO/1518



IRAS ID: 265405

Study Number:

Participant Identification Number for this trial:

## **CONSENT FORM**

| | • | J | valuation of impact on improving the efficier | , , |
|---|---|---|---|---|
| proce | esses and ennancing pation | ent safety in the manag | ement of reactive and spontaneous hypogly | ycaemia. |
| Nam | e of Researcher: Dr Scott | Akker / Dr Craig Stiles | | Please initial box |
| 1.<br>2. | above study. I have had had these answered sati | the opportunity to cons<br>sfactorily. | dated 2.10.2019 (version 1.1) for the ider the information, ask questions and have nonitoring device cannula with transmitter in | |
| | to monitor my glucose le | vels. | | |
| 3. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | | |
| 4. | I understand that relevant sections of my medical notes and data collected during the study may be looked at by individuals from regulatory authorities or from Barts Health NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | | |
| 5. | I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers and Dexcom. | | | |
| 6. | I agree to my General Practitioner being informed of my participation in the study and I agree to my General Practitioner being involved in the study, including any necessary exchange of information about me between my GP and the research team. | | | |
| 7. | I understand that the information held and maintained by Barts Health Trust may be used to help contact me or provide information about my health status. | | | |
| 8. | I agree to take part in the | e above study. | | |
| Name of Participant | | Date | Signature | |
| Name of Person taking consent | | Date | Signature | |